CLINICAL TRIAL: NCT00704548
Title: Antihypertensive Effect of Simvastatin in Hypertensive Patients: a Randomized Clinical Trial With Ambulatory Blood Pressure Monitoring
Brief Title: Antihypertensive Effect of Simvastatin in Hypertensive Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Miguel Gus, Hospital de Clínicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 08014
Record Dates: First submitted 2008-06-23; First posted 2008-06-25 (Estimated); Last update posted 2009-06-26 (Estimated); Status verified 2009-06

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Active Comparator): Simvastatin 40 mg
  Interventions: Drug: Simvastatin 40mg
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Simvastatin 40mg — Simvastatin once daily, orally in the morning period, during eigth weeks
  Arms: 1
Drug: Placebo — Placebo once daily, orally in the morning period, during eigth weeks
  Arms: 2

SUMMARY:
Few trials have investigated the hypotensive effect of the Statins. Most were not specifically aimed at this pleiotropic effect or had methodological problems. The possible hypotensive effect may explain part of the favorable results of the Statins use on cardiovascular prevention independently from its action on the cholesterol profile.

The purpose of this study is to determine the effect of Simvastatin on the blood pressure

DETAILED DESCRIPTION:
This is a randomized double blind parallel clinical trial where hypertensive patients with controlled or uncontrolled blood pressure and without evidence of target-organ damage will be selected. Subjects will receive Simvastatin 40 mg once daily or placebo and a baseline and eight weeks ABPM will performed. The main outcome will be the difference in systolic BP in the 24h-ABPM.

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive patients with controlled or uncontrolled blood pressure

Exclusion Criteria:

* Secondary causes of hypertension;
* Systolic Blood pressure >= 180 mmHg and/or diastolic blood pressure >= 110 mmHg
* Complain of side effects related to Statins
* Diabetes
* Established target-organ damage (myocardial infarction, stroke, angina, heart failure, peripheral vascular disease)
* Renal disease (creatinine > 1,5 mgdl).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-09 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure measured with 24-Ambulatory Blood Pressure Monitoring (24h-ABPM) | Eigth weeks

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Gus, MD, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil